CLINICAL TRIAL: NCT01979627
Title: Safety and Feasibility of Transulnar Artery Approach for Coronary Angiography or Angioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Xianghua (Other)
Responsible Party: Sponsor-Investigator, Fu Xianghua, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fuxhtransulnar
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Intervention; Transulnar; Transradial
Keywords: transulnar approach; transradial approach; angiography; angioplasty

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- transulnar approach group (Experimental): Patients in transulnar group received interventional procedure through ulnar artery
  Interventions: Procedure: transulnar approach interventional procedure
- transradial approach group (Other): patients in transradial group received interventional procedure through radial artery
  Interventions: Procedure: transradial approach interventional procedure

INTERVENTIONS:
Procedure: transulnar approach interventional procedure
  Arms: transulnar approach group
Procedure: transradial approach interventional procedure
  Arms: transradial approach group

SUMMARY:
The transradial approach for coronary angiography and angioplasty is now widely used in catheterization laboratories worldwide, which had been shown as advantages over the conventional femoral and brachial approaches due to the lower incidence of bleeding and other cardiovascular complications. However, the transradial approach does not seem suitable for 5-15% of patients undergoing coronary angiography and angioplasty. The ulnar artery which is one of the two terminal branches of the brachial artery is usually larger than radial artery and it may be as a potential approach for cardiac catheterization. Recently, some reports have demonstrated that the transulnar approach may be both feasible and safe for coronary angiography and angioplasty in selective patients.we performed this study to evaluate the safety and feasibility of transulnar approach coronary catheterization in real world non-selective patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coronary artery disease
* Needed to perform coronary angiography or angioplasty

Exclusion Criteria:

* Arterial circulatory disease in an upper limb
* History of deformity
* Forearm trauma
* Forearm amputated
* Hemodialysis
* Symptomatic peripheral artery disease
* Raynaud's syndrome
* Hemorrhagic disease
* Cardiogenic shock
* Others who were unwilling to participate the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Coronary artery cannulation | 1-12 month
  vascular events including arterial occlusion through ulnar/radial artery approach

SECONDARY OUTCOMES:
Interventional procedure characteristic | during procedure
  The secondary end points included the crossover rate, spasm, total time for the procedure
The access-site related complications | 1-12 month follow up
  The access-site related complications were defined as the occurrence of hematoma, artery stenosis, arteriovenous fistula, pseudoaneurysm, and nerve injury

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Hebei medical university, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Chen J, Huai J, Lin L, Li B, Zhu Y, Yang H. Low-dose aspirin in the prevention of pre-eclampsia in China: postpartum hemorrhage in subgroups of women according to their characteristics and potential bleeding risk. Chin Med J (Engl). 2023 Mar 5;136(5):550-555. doi: 10.1097/CM9.0000000000002545. PMID 36914957
- [Derived] Liu L, Xu XT, Yu Y, Sun Q, Yang Y, Qiu HB. Neural control of pressure support ventilation improved patient-ventilator synchrony in patients with different respiratory system mechanical properties: a prospective, crossover trial. Chin Med J (Engl). 2021 Jan 19;134(3):281-291. doi: 10.1097/CM9.0000000000001357. PMID 33470654
- [Derived] Bi X, Wang Q, Liu D, Gan Q, Liu L. Is the Complication Rate of Ulnar and Radial Approaches for Coronary Artery Intervention the Same? Angiology. 2017 Nov;68(10):919-925. doi: 10.1177/0003319717703226. Epub 2017 Apr 7. PMID 28387125
- [Derived] Bi XL, Fu XH, Gu XS, Wang YB, Li W, Wei LY, Fan YM, Bai SR. Influence of Puncture Site on Radial Artery Occlusion After Transradial Coronary Intervention. Chin Med J (Engl). 2016 Apr 20;129(8):898-902. doi: 10.4103/0366-6999.179795. PMID 27064032